CLINICAL TRIAL: NCT04898998
Title: TENS to Alleviate the Effect of Xerostomia (Dry Mouth) After Surgery
Brief Title: TENS to Alleviate the Effect of Thirty After Surgery Xerostomia (Dry Mouth) After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiu-Ling Yang, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901244A3C501
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Complications
Keywords: postoperative thirty, postoperative recovery room, complain
MeSH Terms: conditions — Postoperative Complications | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS to alleviate the effect of thirsty after surgery (Experimental): Transcutaneous electrical nerve stimulation (TENS) on experimental group 20 mins to treatment postoperative thirsty.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Routine care to alleviate the effect of xerostomia (dry mouth) after surgery (Placebo Comparator): routine care
  Interventions: Other: routine care

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Surgical patients under general anesthesia were recruited from a medical center. Each patient was randomly assigned to the experimental group (TENS) or control group (routine care).
  Arms: TENS to alleviate the effect of thirsty after surgery
Other: routine care — routine care
  Arms: Routine care to alleviate the effect of xerostomia (dry mouth) after surgery

SUMMARY:
Dry mouth of postoperative makes the patient feel thirst, and the pain of the lips is cracked. It will also make the sputum thick and sticky, making it difficult for the patient to cough by himself. Especially the elderly may have sputum accumulation and pneumonia. Dry mouth can easily change the pH value in the mouth, destroy the environment in the mouth, and increase the chance of oral mucosal lesions, ulcers and infections. The physical discomfort can lead to psychological effects such as anxiety, irritability, and irritability. The incidence of dry mouth was 88%, 6-8 hours after abdominal surgery. Although the incidence is high, compared with other complications after surgery (such as: pain, bleeding, etc.), dry mouth after surgery is less important, and is underestimated, unmeasured, unrecorded and untreated. Initiating the motivation of this study, it is hoped that through research to understand the relevant factors causing dry mouth after surgery, and using transcutaneous electrical nerve stimulation (TENS) to improve the symptoms of dry mouth after surgery. The first phase is to describe the relevant studies with the aim of understanding the relevant factors that contribute to dry mouth after surgery. This study will understand and pay attention to the post-operative dry mouth. It is hoped that through this study, the problem of dry mouth after surgery will be improved, and the comfort of the recovery period after surgery will be improved, so that patients can get better care and promote the quality of care.

DETAILED DESCRIPTION:
Introduction A postoperative thirst is one of the major complaints in the recovery room. The purpose of this experimental study was to compare the efficiency of reducing postoperative thirst by transcutaneous electrical nerve stimulation (TENS) and routine care.

Methods Surgical patients under general anesthesia were recruited from a medical center. Each patient was randomly assigned to the experimental group (TENS) or control group (routine care). Experimental group had 53 patients and control group had 52 patients fitted in the inclusion and exclusion criteria and completed data collection. The intensity of thirst was measured pretreatment, immediately after treatment and 30 minutes after treatment. All data were managed by SPSS for Windows (version 21.0). Descriptive and inferential statistics (Chi-square test, t-test, generalized estimating equation regression analysis) were performed to identify the relationships that were proposed.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology (ASA) physical status I-ΙII, elective abdominal surgery, >20 years old

Exclusion Criteria:

* pregnancy, epilepsy, unconscious

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The intModified Schirmer tear strip Test measured intensity of thirst | up to 30 minutes
  Change from Baseline intensity of thirst was measured pre-treatment, immediately after treatment and 30 minutes after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hsiu-Ling Yang, Taoyuan District, Fuxing St., Guishan Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No